CLINICAL TRIAL: NCT04053621
Title: Pirofosfato de Tiamina Como Coadyuvante de la Metformina en el Tratamiento de Pacientes Con Diabetes Mellitus Tipo 2
Brief Title: Co-administration of Thiamine Pyrophosphate and Metformin in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorios Manuell SA (Industry)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Dr. Melchor Alpízar Salazar, Principal investigator, Laboratorios Manuell SA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2336732
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: metformin; thiamine pyrophosphate; B1 vitamin; type 2 diabetes mellitus; metabolic pathways
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Thiamine Pyrophosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Metformin at patient´s tolerated oral dose (maximum of 2550 mg per day) and thiamine pyrophosphate (weekly dose of 1 gram administered by IV: 25 ml of thiamine pyrophosphate + 250 ml saline solution at a 60-80 drops/minute rate).
  Total duration of 12 weeks.
  Interventions: Dietary Supplement: Thiamine pyrophosphate; Drug: Metformin
- Placebo group (Placebo Comparator): Metformin at patient´s tolerated oral dose (maximum of 2550 mg per day) and weekly administration of 275 ml of saline solution at a 60-80 drops/minute rate).
  Total duration of 12 weeks.
  Interventions: Other: Placebo; Drug: Metformin

INTERVENTIONS:
Dietary Supplement: Thiamine pyrophosphate — 12 weeks of weekly dose of 1 gram of thiamine pyrophosphate administered in an intravenous manner with saline solution
  Other Names: Cocarboxylase
  Arms: Experimental group
Other: Placebo — 12 weeks of weekly dose of 275 ml of saline solution administered in an intravenous manner
  Arms: Placebo group
Drug: Metformin — All participants will continue taking metformin in their previous established tolerated dose for the duration of the study

SUMMARY:
Chronic non-infectious diseases have a bigger impact and a higher prevalence every day world-wide. Among them, diabetes stands out being the number one cause of death from degenerative chronic illness in Mexico. Diabetes not only affects quality of life, it can also lead to severe complications that have a great economic impact as well as a health impact on the patient and their family. Some of the complications include liver failure and hypertension. This whole problem can be dated back to an initial hyperglycemic state that when left untreated further develops into insulin resistance, chronic inflammation, metabolic syndrome and diabetes. The purpose of this study is to stop this chain reaction that starts with every hyperglycemic patient by adding thiamine pyrophosphate to the treatment plan of patients diagnosed with type 2 diabetes that are poorly managed with metformin monotherapy. Thiamine pyrophosphate is a form of B1 vitamin that plays an important role as a coenzyme in multiple metabolic routes including the link between glycolysis and Krebs cycle, fatty acids metabolism and branched-chain amino acid metabolism. By doing so, these pathways improve their function and efficiency and thereby utilize plasma glucose. This in turn, decreases the formation of advanced glycation end products (AGEs) which prevents the formation of reactive oxygen and nitrogen species, ultimately there is also an anti-oxidative mechanism involved that improves the inflammatory state the patient is living with. Our hypothesis is that by adding thiamine pyrophosphate to the treatment of patients taking metformin, there will be important progress regarding the inflammatory and metabolic control of patients with type 2 diabetes.

The study will have a duration of approximately 4 months after the total sample is recruited. During this time, subjects will first be examined to determine their eligibility according to the pre-established criteria, in case of inclusion in the study they will sign an informed consent after reading it thoroughly and having answered all their questions. Baseline labs will be taken for every subject for future comparison. They will then be randomized into two parallel groups: an experimental group that will receive weekly infusions of saline infused with 1 gram of thiamine pyrophosphate or a placebo group that will also receive weekly infusions of pure saline. The patients as well as the doctors treating them will be blinded to the assignment of either group. This model will be carried out for a duration of 12 weeks total, during which every patient will continue their metformin treatment with their tolerated dose. There will be verification of treatment adherence by counting the metformin pills during every weekly visit. For the assessment of dependent variables there will be a visit every month with a blinded doctor. These visits will be for: physical and clinical evaluation, evaluation of adverse events, evaluation of treatment adherence and a heart rate variability study. The first and third months a questionnaire about lifestyle will be added to the visit schedule. On the third month, final lab tests will be performed. Finally, one month after completing the treatment, a final visit will be scheduled for a clinical and physical evaluation to make sure there are no problems.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosed type 2 diabetes mellitus
* HbA1c between 7.5 and 11%
* monotherapy treatment with metformin at tolerated successful dose

Exclusion Criteria:

* glomerular filtration rate <60 ml/min/1.73m2
* cardiac o respiratory insufficiency
* liver enzymes 3 times higher than normal parameters
* known allergy to metformin or thiamine pyrophosphate
* pregnancy, lactation or fertile age without a contraceptive method
* participation in another study in the last 6 months
* programmed surgery for the next 4 months
* treatment with any other hypoglycemic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
hemoglobin A1c | Change from baseline at 3 months
  percentage

SECONDARY OUTCOMES:
fasting plasma glucose | Change from baseline at 3 months
  mg/dl
Lipids profile | Change from baseline at 3 months
  Concentration of total cholesterol, HDL, LDL and triglycerides (mg/dl)
inflammation markers | Change from baseline at 3 months
  Concentration of PCR, IL-6, TNF-alpha, nitric oxyde, superoxide dismutase, free fatty acids, catalase
Lifestyle measurement | Change from baseline at 3 months
  IMEVID questionnaire (instrumento para medir el estilo de vida en diabéticos). Total scores are reported from 0-100. Higher scores are associated with a better lifestyle, >75 quartile is considered a good score.
heart rate variability | Change from baseline at 3 months
  measured in milliseconds
arterial elasticity | Change from baseline at 3 months
  Using the HDI/PulseWave instrument

CONTACTS AND LOCATIONS:
Overall Officials: Melchor Alpizar, MD, PhD, Principal Investigator — Centro Especializado en Diabetes, Obesidad, Prevención y Enfermedades Cardiovasculares, S.C.
Locations (1):
- Centro Especializado en Diabetes, Obesidad, Prevención y Enfermedades Cardiovasculares, S.C., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alaei Shahmiri F, Soares MJ, Zhao Y, Sherriff J. High-dose thiamine supplementation improves glucose tolerance in hyperglycemic individuals: a randomized, double-blind cross-over trial. Eur J Nutr. 2013 Oct;52(7):1821-4. doi: 10.1007/s00394-013-0534-6. Epub 2013 May 29. PMID 23715873
- [Background] Al-Daghri NM, Alharbi M, Wani K, Abd-Alrahman SH, Sheshah E, Alokail MS. Biochemical changes correlated with blood thiamine and its phosphate esters levels in patients with diabetes type 1 (DMT1). Int J Clin Exp Pathol. 2015 Oct 1;8(10):13483-8. eCollection 2015. PMID 26722561
- [Background] Benítez-Rodríguez MT. Actualidades del Pirofosfato de Tiamina o Carboxilasa. 1st ed. México: Litográfica Santander; 2013.
- [Background] Elksnis A, Martinell M, Eriksson O, Espes D. Heterogeneity of Metabolic Defects in Type 2 Diabetes and Its Relation to Reactive Oxygen Species and Alterations in Beta-Cell Mass. Front Physiol. 2019 Feb 13;10:107. doi: 10.3389/fphys.2019.00107. eCollection 2019. PMID 30837889
- [Background] Lopez-Carmona JM, Rodriguez-Moctezuma JR, Ariza-Andraca CR, Martinez-Bermudez M. [Lifestyle and metabolic control in patients with type 2 diabetes mellitus. Construct validation of IMEVID questionnaire]. Aten Primaria. 2004 Jan;33(1):20-7. doi: 10.1016/s0212-6567(04)78873-3. Spanish. PMID 14746741
- [Background] Pacal L, Kuricova K, Kankova K. Evidence for altered thiamine metabolism in diabetes: Is there a potential to oppose gluco- and lipotoxicity by rational supplementation? World J Diabetes. 2014 Jun 15;5(3):288-95. doi: 10.4239/wjd.v5.i3.288. PMID 24936250
- [Background] Shapoval GS, Babii LV, Kruglyak OS, Vovk AI. Antioxidant activity of thiamine and its structural analogs in reactions with electrochemically generated hydroxyl radicals and hydrogen peroxide. Theor Exp Chem. 2011; 47, 1: 55 - 60.